CLINICAL TRIAL: NCT01059032
Title: Enhancement and Restoring of Low Dose Abdominal CT Images by a Novel Adaptive Nonlinear 3D Post Processing Filter - a Prospective Blinded Interventional Study
Brief Title: Enhancement and Restoring of Low Dose Abdominal CT Images
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lars Borgen (Other)
Collaborators: Sykehuset Buskerud HF (Other)
Responsible Party: Sponsor-Investigator, Lars Borgen, MD, University of Oslo
Organization: University of Oslo (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 15017044793
Record Dates: First submitted 2010-01-21; First posted 2010-01-29 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2009-11

CONDITIONS: Radiation Protection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Unenhanced images (No Intervention)
- Enhanced images (Other): Enhanced images
  Interventions: Other: Using a 3 dimentional post processing filter

INTERVENTIONS:
Other: Using a 3 dimentional post processing filter — Using a 3 dimentional post processing filter
  Arms: Enhanced images

SUMMARY:
Through the rapid growth of multislice Computer Tomography (CT) imaging, radiation protection has become a major issue in the radiological community. Optimizing CT scanning is a key task when keeping the radiation doses as low as reasonable achievable (the ALARA principle). Post processing filters can improve and restore grainy and noisy low dose CT images by enhancing structure and reducing image noise. In our study of 10 patients, the investigators perform a preliminary evaluation of a novel post processing filter, which does picture element correlations in all three spatial dimensions. By comparing normal dose pictures with unprocessed low-dose pictures and pictures processed with two dimentional (2D) and three dimentional (3D) filters,the investigators will be able to assess the possible clinical value of the 3D filter. This project is collaboration between Buskerud Hospital (BU), Buskerud University College, Norwegian Radiation Protection Authority (NRPA) and Center for Medical Image Science and Visualization (CMIV). The project is part of the PhD of Lars Borgen.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients, Male or female,Age above 60 years, Referred to our department for an abdominal CT with intravenous contrast.

Exclusion Criteria:

* Abdominal diameter less than 80cm or larger than 100cm, Gross pancreatic pathology, Gross anatomic anomalies in the investigated region, Intolerance of intravenous contrast

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-12; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Rating of image quality | 3-6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Buskerud Hospital, Drammen, Norway